CLINICAL TRIAL: NCT06584331
Title: HEMODYNAMIC and BIOCHEMICAL RESPONSES to 10 DAYS of BEETROOT JUICE INTAKE in POSTMENOPAUSAL HYPERTENSIVE WOMEN
Brief Title: BEETROOT JUICE INTAKE in POSTMENOPAUSAL HYPERTENSIVE WOMEN
Acronym: EBJIPHW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Ana Luiza Amaral Ribeiro, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01.78649524.4.0000.5152; APQ-01874-18 (Other Grant/Funding Number: FAPEMIG); 175522/2023-5 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2024-08-26; First posted 2024-09-04 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Menopause
Keywords: beetroot juice; hypertension; postmenopausal; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 dose of beetroot juice (Experimental): The volunteers will ingest 70 ml of beetroot juice with 400 mg of nitrate every morning for 10 days
  Interventions: Dietary Supplement: 1 dose of Beetroot juice intake
- 2 doses of beetroot juice (Experimental): This group will ingest 2 shots of 70 ml of beetroot juice with 400mg of nitrate, in each shot, for 10 days.
  Interventions: Dietary Supplement: 2 doses of Beetroot juice intake
- Placebo (Placebo Comparator): In this group, the participants will receive a low-nitrate beetroot juice dose to consume in the morning.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 1 dose of Beetroot juice intake — The volunteers will ingest 70 ml of beetroot juice with 400 mg of nitrate every morning for 10 days
  Arms: 1 dose of beetroot juice
Dietary Supplement: 2 doses of Beetroot juice intake — This group will ingest 2 shots of 70 ml of beetroot juice with 400mg of nitrate, in each shot, for 10 days.
  Arms: 2 doses of beetroot juice
Dietary Supplement: Placebo — In this group, the participants will receive 70ml of low-nitrate beetroot juice to consume in the morning.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to verify the hemodynamic and biomarker responses of beetroot juice intake in postmenopausal women with hypertension. The main questions it aims to answer are:

Is beetroot juice dose related to better hemodynamic responses in hypertensive postmenopausal women? Is beetroot juice dose related to better oxidative stress profile responses in hypertensive postmenopausal women?

The investigators will conduct a parallel clinical study with 10 days of intervention, in which 48 women will be randomized into 3 groups: 1) Two shots of beetroot juice intake per day (800mg of NO3-); 2) One shot of beetroot juice intake per day (400mg of NO3-); 3) placebo intake (beetroot juice without NO3-).

DETAILED DESCRIPTION:
The entire intervention will take place at the Physical Education campus of University, in the Cardiorespiratory and Metabolic Physiology Laboratory (LAFICAM). The recruitment and approach of the volunteers will occur through media dissemination, such as radio announcements, television programs, and social media through digital media. After the dissemination, volunteers will make contact via phone, email, or social media, and a preliminary registration will take place. After this registration, the researchers will verify which volunteers meet the inclusion criteria, and only then will the recruitment take place.

The volunteers will be invited to come to LAFICAM to be informed about the intervention program and then sign the informed consent form. Before starting the intervention program, all volunteers must present a medical certificate clearing them to participate in a physical exercise training program; once the certificate is submitted, initial tests and general evaluations will be conducted.

The initial evaluations will consist of a questionnaire, anthropometric and body composition assessment, and evaluation of the physical activity level. After the questionnaires are administered, a familiarization with the sensory perceptions of beetroot juice will be conducted. This familiarization is important to verify if the volunteers are fit to carry out the intervention.

The volunteers will be randomized into three groups: Group 1: the volunteers will ingest two shots containing 70 ml of beetroot juice with 400 mg of nitrate per day, one shot in the mornig and one shot at night, for 10 days; Group 2: this group will intake 70 ml of beetroot juice with 400 mg of nitrate every morning.

Group 3: this group will intake 70 ml of beetroot juice without nitrate for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Amenorrhea for at least 12 months
* Controlled hypertension

Exclusion Criteria:

* Decompensated hypertension in stages 2 and 3
* Having a history of stroke or acute myocardial infarction
* Smoker
* Having a diagnosis of Diabetes Mellitus
* Using hormone therapy.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 11 days
  Volunteers will undergo blood pressure tests at the beginning, in the middle and after the 10 days of intervention. To assess blood pressure (BP), researchers will use the Dyna Mapa + Cardius® device, programmed with measurements to be taken every 20 min. Together with this device, the volunteers filled out a daily record of activities such as sleep, work, food, or any event that could interfere with BP or measurements. In a standardized manner, the device was set at 7 a.m., and measurements were considered valid when 24h of monitoring were obtained. Resting BP was measured with the same device after 15 min of rest in a sitting position, and for the analysis of the pressure curve, time 0 was adopted when the monitor was placed. Sytolic BP, diastolic BP, and mean BP in periods of awake, sleep and 24 h were analyzed.

SECONDARY OUTCOMES:
Stroop color and word test | 11 days
  The evaluation of the blood pressure (BP) reactivity was carried out under mental stress, through the electronic version of Stroop protocol (3 minutes). For the test, the volunteers sited in front of a computer screen with a headset and listened to a voice speaking names of different colors and with images changing every 2 seconds. Each image consisted of a word forming the name of a color, with the word's letters color being different from the color's name, and with the bottom of the word with another color different from the color of the word and the color's name formed by the word. The volunteers should speak as quickly as possible the name of the color formed by the letters in the image. Before the test, baseline BP were measure once after resting in siting position during 15 minutes. During the test, the volunteers BP was measured every minute, through the auscultatory method.
Heart rate variability | 11 days
  Resting R-R intervals will be recorded for 15 min in the seated position using an HR monitor (POLAR® RS800cx; Polar Electro Oy, Finland; sampling frequency = 1000 Hz) with spontaneous breathing. Data will be downloaded to a computer using an infrared interface with specific software (POLAR PRO TRAINER5®, Polar Electro, Kempele, Finland). Heart rate variability (HRV) analysis was performed using KUBIOS HRV 3.0. Prior to the analysis, the signal will be visually inspected and filtered, and a range of 5 min interval with few artifacts will be selected near the end of the recording for analysis. The resulting R-R intervals will be analyzed in the time domain, in the frequency domain using spectral analysis (Fast Fourier Transform), and non-linearly through the Poincaré diagram.
Superoxide Dismutase | 11 days
  Superoxide Dismutase (SOD) activity will be assessed by inhibition of pyrogallol autoxidation. Samples will be mixed with 50 mmol L Tris-HCl buffer (pH 8.2) containing 1 mmol L EDTA to deactivate metal-dependent enzymes, 80 U mL 1 catalase, and 24 mmol L 1 pyrogallol, and the kinetic assay will be monitored for 10 min at 420 nm using an analytical curve constructed with SOD as a standard.
Catalase | 11 days
  Catalase (CAT) activity will be based on the decomposition of hydrogen peroxide. Samples will be mixed with a 10 mmol_L^-1 potassium phosphate buffer (pH 7.0 containing 0.2% hydrogen peroxide. Hydrogen peroxide decomposition will be monitored at 240 nm for 10 min.
Glutathione Peroxidase | 11 days
  To measure glutathione peroxidase (GPx) activity, plasma will be incubated with GPx buffer (100 mM potassium phosphate containing 1 mM EDTA, pH 7.7), sodium azide (40 mM), glutathione (GSH) (diluted in 5% metaphosphoric acid), glutathione reductase (GR) (diluted in GPx buffer), NADPH (diluted with 5% sodium bicarbonate), and tert-butyl hydroperoxide (0.5 mM). The reduction in NADPH concentration will be assessed for 10 min in a spectrophotometer at 340 nm.
Total antioxidant capacity due to ferric-reducing antioxidant power (FRAP) | 11 days
  The total antioxidant capacity due to iron reducing antioxidant power (FRAP) will be determined by the ability of the antioxidants present in the blood samples to reduce Fe3+ to Fe2+, which is chelated by TPTZ (2,4,6-tris(2-pyridyl)-s-triazine) and forms the Fe2+ TPTZ complex. This complex will be quantified in a spectrophotometer at 593 nm, and the antioxidant activity will be determined by means of an analytical curve, constructed with trolox as a standard.
Reduced glutathione (GSH) | 11 days
  Plasma proteins will be precipitated with metaphosphoric acid (MPA) and centrifuged at 7000 g for 10 min. The supernatant will be collected and mixed with 100 mM sodium phosphate buffer (pH 8.0) containing 5 mM EDTA and 15 μL ortho-phthaldialdehyde (1 mg/mL in methanol, HPLC grade, 99.9%). The solution will be incubated in the dark at room temperature for 15 min. Fluorescence will be read at 350 nm (excitation) and 420 nm (emission). Glutathione (GSH) concentrations of the sample will be calculated using a GSH standard curve (0.001-0.1 mM)
Human cytokines | 11 days
  Human cytokines (IL-8, IL-1β, IL-6, TNF, IL-10 and IL-12p70) in serum samples will be measured by flow cytometry technique (FACSCantoII BD™, San Jose, CA, USA) using a human inflammatory cytokine kit (BD™ Cytometric Bead Array (CBA), BD Biosciences, San Jose, CA, USA) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- FAEFI, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
The IPD will not be made available, but it can be sent by email upon request.